CLINICAL TRIAL: NCT01603875
Title: Immune Response in Adults to Pre-exposure Rabies Vaccination and Simulated Post-exposure Rabies Booster Vaccination With a New Chromatographically Purified Vero-cell Rabies Vaccine(SPEEDA®) : a Randomized Controlled Trial With Purified Vero-cell Rabies Vaccine (PVRV)
Brief Title: Immune Response in Adults to PrEP and Simulated Booster PEP With a New CPRV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Saovabha Memorial Institute (Other)
Responsible Party: Principal Investigator, Jaruboot Angsanakul, MD, Jaruboot Angsanakul, Medical Officer 4, Queen Saovabha Memorial Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC5506
Record Dates: First submitted 2012-05-16; First posted 2012-05-23 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-01

CONDITIONS: Efficacy of the New CPRV
Keywords: CPRV; SPEEDA; intradermal; pre-exposure; booster

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PrEP and Simulated PEP with PVRV by intramuscular route (Active Comparator)
  Interventions: Biological: New Chromatographically Purified Vero-cell Rabies vaccine(new CPRV).
- PrEP and Simulated PEP with new CPRV by intramuscular route (Experimental)
  Interventions: Biological: New Chromatographically Purified Vero-cell Rabies vaccine(new CPRV).
- PrEP and Simulated PEP with new CPRV by intradermal route (Experimental)
  Interventions: Biological: New Chromatographically Purified Vero-cell Rabies vaccine(new CPRV).

INTERVENTIONS:
Biological: New Chromatographically Purified Vero-cell Rabies vaccine(new CPRV). — new CPRV 0.1 ml intradermal route and 0.5 ml intramuscular route are the experimental intervention

SUMMARY:
Pre exposure rabies vaccination with a new Chromatographically Purified Vero-cell Rabies Vaccine(SPEEDA) is as effective as Purified Vero-cell Rabies vaccine.

After the pre exposure rabies vaccination with a new Chromatographically Purified Vero-cell Rabies Vaccine(SPEEDA), the Rabies neutralizing antibodies in all patients on day 42 are 0.5 IU/ml or more.

And Simulated post-exposure rabies booster vaccination with a new Chromatographically Purified Vero-cell Rabies Vaccine(SPEEDA) is as effective as Purified Vero-cell Rabies vaccine.

After the simulated post-exposure rabies booster vaccination with a new Chromatographically Purified Vero-cell Rabies Vaccine(SPEEDA), the Rabies neutralizing antibodies in all patients on day 14 after the booster are 0.5 IU/ml or more.

DETAILED DESCRIPTION:
Pre-exposure vaccination will be done according to standard protocol. Participants will be injected with one dose on day 0, 7 and 28. Blood samples will be taken on day 0, 28 and 42 after the first vaccination dose.

360 days later, participants will receive simulated post-exposure rabies booster vaccination one dose on day 0 and 3. Blood samples will be taken again on day 0(360 days) and 14(374 days) after the booster vaccination.

Rabies neutralizing antibody levels will be measured by Rapid Fluorescent Focus Inhibition Test(RFFIT). And the levels of 0.5 IU/ml or more is considered acceptable protective level.

For statistical analysis, percentage of subjects achieving seroconversion (defined as RNab ≥ 0.5 IU/ mL) are determine at each sampling time. The average of the titer used in this study is Geometric mean titer(GMT). 95 percent confidence interval(95% CI) of the GMT will be calculated for each study group from individual measurements of serum rabies antibody levels at each sampling time. One-way ANOVA would be used to calculated the significance of the difference between the GMT of three groups, SPEEDA® intradermal injection, SPEEDA® intramuscular injection and PVRV intramuscular injection. The primary criterion for this comparison are the rabies antibody value on day 42 (2 weeks after the third vaccine dose of pre-exposure vaccination) and on day 374(2 weeks after the first vaccine dose of booster vaccination). Results will be deemed statistically significant at p < 0.05. Safety data (immediate, local and systemic reactions) were summarized as numbers and percentages.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Can visit according to the protocol

Exclusion Criteria:

* Fever
* Acute illness
* History of rabies vaccination
* Allergic to the vaccines' component
* Immunosuppressive conditions such as HIV infection, transplantation, chronic renal failure, received steroid or immunosuppressive drugs and anti-malarial drugs within previous two months or any blood products within previous three months
* Female participant must not be pregnant
* All female participant must have urine pregnancy test negative prior to participate the study

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terapong Tantawichien, M.D., Principal Investigator — Queen Saovabha Memorial Institute
Locations (1):
- Queen Saovabha Memorial Institute, Bangkok, Bangkok, Thailand

REFERENCES:
- See also: Contact information — http://www.saovabha.com/en/contactus.asp

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 66 subjects from Faculty of Veterinarian, Chulalongkorn University. The recruitment held between June 25, 2012 and July 2, 2012. Others 39 subjects was recruited from Faculty of Veterinarian, Mahanakorn University of Technology.
Period: Overall Study
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route
Started | 35 | 35 | 35
Completed | 28 | 27 | 26
Not Completed | 7 | 8 | 9
Not completed — Preexisting rabies antibody | 3 | 4 | 3
Not completed — Lost to Follow-up | 4 | 3 | 6
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route | Total
Number analyzed (Participants) | 28 | 27 | 26 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.96 (1.138) | 20.04 (5.633) | 18.92 (0.744) | 19.31 (3.345)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 19 | 59
  Male | 6 | 9 | 7 | 22
Region of Enrollment [Number; unit: participants]
  Thailand | 28 | 27 | 26 | 81

OUTCOME MEASURES:

1. Primary Outcome: Rabies Neutralizing Antibodies Determine by Rapid Fluorescent Focus Inhibition Test (RFFIT)
Description: Blood samples will be drawn on day 0(After the first injection). The samples will be centrifuged and kept as serum under - 20 degree Celsius. The serum will be test by Rapid Florescent Focus Inhibition Test. Rabies neutralizing antibody levels will be determined and expressed in international units per mL. Percentage of Subjects achieving seroconversion (defined as RNab ≥ 0.5 IU/ mL) are determine at each sampling time.
Time Frame: on day 0
Measure: Geometric Mean (Full Range); unit: International unit per ml
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route
Number analyzed (Participants) | 31 | 31 | 32
International unit per ml | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Rabies Neutralizing Antibodies Determine by Rapid Fluorescent Focus Inhibition Test (RFFIT)
Description: Blood samples will be drawn on day 28(After the first injection). The samples will be centrifuged and kept as serum under - 20 degree Celsius. The serum will be test by Rapid Florescent Focus Inhibition Test. Rabies neutralizing antibody levels will be determined and expressed in international units per mL. Percentage of Subjects achieving seroconversion (defined as RNab ≥ 0.5 IU/ mL) are determine at each sampling time.
Time Frame: on day 28
Measure: Geometric Mean (Full Range); unit: International unit per ml
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route
Number analyzed (Participants) | 31 | 31 | 32
International unit per ml | 2.67 [0.57 to 11.81] | 4.23 [0.46 to 19.03] | 1.83 [0.16 to 17.45]

3. Primary Outcome: Rabies Neutralizing Antibodies Determine by Rapid Fluorescent Focus Inhibition Test (RFFIT)
Description: Blood samples will be drawn on day 42(After the first injection). The samples will be centrifuged and kept as serum under - 20 degree Celsius. The serum will be test by Rapid Florescent Focus Inhibition Test. Rabies neutralizing antibody levels will be determined and expressed in international units per mL. Percentage of Subjects achieving seroconversion (defined as RNab ≥ 0.5 IU/ mL) are determine at each sampling time.
Time Frame: on day 42
Measure: Geometric Mean (Full Range); unit: International unit per ml
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route
Number analyzed (Participants) | 31 | 31 | 32
International unit per ml | 11.49 [2.38 to 51.54] | 14.23 [1.83 to 64.00] | 5.02 [0.59 to 26.91]

4. Primary Outcome: Rabies Neutralizing Antibodies Determine by Rapid Fluorescent Focus Inhibition Test (RFFIT)
Description: Blood samples will be drawn on day 360(After the first injection). The samples will be centrifuged and kept as serum under - 20 degree Celsius. The serum will be test by Rapid Florescent Focus Inhibition Test. Rabies neutralizing antibody levels will be determined and expressed in international units per mL. Percentage of Subjects achieving seroconversion (defined as RNab ≥ 0.5 IU/ mL) are determine at each sampling time.
Time Frame: on day 360
Measure: Geometric Mean (Full Range); unit: International unit per ml
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route
Number analyzed (Participants) | 28 | 27 | 26
International unit per ml | 0.55 [0.16 to 1.83] | 0.64 [0.13 to 3.67] | 0.28 [0.07 to 1.19]

5. Primary Outcome: Rabies Neutralizing Antibodies Determine by Rapid Fluorescent Focus Inhibition Test (RFFIT)
Description: Blood samples will be drawn on day 374(After the first injection). The samples will be centrifuged and kept as serum under - 20 degree Celsius. The serum will be test by Rapid Florescent Focus Inhibition Test. Rabies neutralizing antibody levels will be determined and expressed in international units per mL. Percentage of Subjects achieving seroconversion (defined as RNab ≥ 0.5 IU/ mL) are determine at each sampling time.
Time Frame: on day 374
Measure: Geometric Mean (Full Range); unit: International unit per ml
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route
Number analyzed (Participants) | 28 | 27 | 26
International unit per ml | 29.16 [7.66 to 112.40] | 45.99 [4.36 to 693.38] | 11.93 [3.22 to 66.83]

6. Secondary Outcome: Side Effects of the Vaccines. These Include Pain, Swelling, Redness, Myalgia, Rash, Fever. Serious Adverse Events Will Also be Recorded.
Description: There are five injections, on day 0, 7, 28, 360 and 363.
  The side effects will be record in number and percentage.
Time Frame: up to 7 days after each injection
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 42 days since the first dose was administered. One year later, 14 days since the first booster dose was administered.
Description: Pain, pruritus, erythema, induration, fever, urticaria, arthralgia, myalgia, dizziness, headache, nausea, vomiting, lymphadenopathy were recorded.
Arm/Group | PrEP and Simulated PEP With PVRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intramuscular Route | PrEP and Simulated PEP With New CPRV by Intradermal Route
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 35/35 | 35/35 | 35/35
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrEP and Simulated PEP With PVRV by Intramuscular Route (N=35) | PrEP and Simulated PEP With New CPRV by Intramuscular Route (N=35) | PrEP and Simulated PEP With New CPRV by Intradermal Route (N=35)
pain (Injury, poisoning and procedural complications) | 28 (149) | 27 (147) | 15 (148)
pruritus (Skin and subcutaneous tissue disorders) | 5 (7) | 6 (8) | 16 (38)
erythema (Skin and subcutaneous tissue disorders) | 4 | 1 | 26
induration (Skin and subcutaneous tissue disorders) | 2 | 1 | 26
fever (General disorders) | 8 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No